CLINICAL TRIAL: NCT00302419
Title: Effect of Complementary Intracoronary Streptokinase Administration Immediately After Primary Percutaneous Coronary Intervention on Microvascular Perfusion and Late Term Infarct Size in Patients With Acute Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Istanbul University Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5737
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; primary angioplasty; streptokinase; microvasculature
MeSH Terms: interventions — Streptokinase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Following standard primary percutaneous coronary intervention for ST elevation acute myocardial infarction 250.000 U intracoronary Streptokinase will be given
  Interventions: Drug: intracoronary infusion,; Procedure: primary percutaneous coronary angioplasty
- 2 (Active Comparator): Standard percutaneous coronary intervention for ST elevation myocardial infarction will be performed
  Interventions: Procedure: primary percutaneous coronary angioplasty

INTERVENTIONS:
Drug: intracoronary infusion, — streptokinase, 250,000 units
  Other Names: Streptase
  Arms: 1
Procedure: primary percutaneous coronary angioplasty

SUMMARY:
The investigators hypothesized that complementary intracoronary streptokinase administration to primary percutaneous intervention in patients with acute myocardial infarction may provide further improvement in myocardial perfusion by dissolving microvascular thrombus [in situ formed or embolized from proximal site (spontaneous or following PCI)] and fibrin.

DETAILED DESCRIPTION:
Mechanical reperfusion for acute myocardial infarction (AMI) targets optimal revascularization of the epicardial artery but also aims at improved myocardial salvage. The goal of reperfusion therapies has shifted to include reperfusion downstream at the level of capillary bed, and it might be more appropriate that the hypothesis now be termed "the time dependent open artery and open microvascular hypothesis." Failure to achieve myocardial reperfusion despite the presence of a patent coronary artery has been termed the "no-reflow" phenomenon and attributed to microvascular dysfunction. It has become apparent that clinical outcomes are not only associated with patency of the epicardial artery, but also with patency of the microcirculation. Persistent impairment of microcirculation is associated with poor clinical outcome. Complete reperfusion in AMI settings necessitates reopening of the all consecutive vascular compartments all the way through the coronary circulation. But, embolization following percutaneous coronary intervention (PCI) and in situ microthrombi generation at the microvascular level makes this goal difficult to achieve. For this reason, mechanical intervention to the epicardial coronary artery with or without using distal protection wouldn't be enough to achieve ideal reperfusion at the ultimate (microvascular) level. At this point, it has become more evident that we need to develop more competent and feasible reperfusion strategies which can help us to achieve reperfusion as complete as possible at all levels.

Hypothesis:

Complementary intracoronary streptokinase administration to primary PCI may provide further improvement in myocardial perfusion by dissolving microvascular thrombus [in situ formed or embolized from proximal site (spontaneous or following PCI)] and fibrin. Improvement in microvascular perfusion may translate into reduction in infarct size and improvement in left ventricular function at long term.

ELIGIBILITY:
Inclusion criteria:

* Continuous chest pain that lasted > 30 minutes within the preceding 12 hours
* ST-segment elevation of at least 1 mm in 2 contiguous leads on the 12 leads ECG
* Infarct related artery (IRA) occlusion (TIMI grade 0) at the angiography
* Angiographically detected culprit coronary artery lesion deemed suitable for PCI

Exclusion Criteria:

* Contraindications to streptokinase, tirofiban, aspirin, clopidogrel, or heparin
* Culprit lesion in saphenous vein graft
* TIMI grade II-III flow in IRA
* Additional epicardial stenosis in the IRA distal to stented segment (significant or insignificant)
* Presence of left bundle branch block
* History of prior MI
* Mechanical ventilation or inotropic support

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2004-10; Primary Completion 2006-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Primary end points defined as the indices of the microvascular perfusion which is going to be assessed on day 2 (48 hours after the primary PCI)and infarct size at 6 months. | 6 months
Index of microvascular resistance, | 48 hours
Coronary flow reserve | 48 hours
Left ventricular infarct size by SPECT at six months. | 6 months

SECONDARY OUTCOMES:
Death | 1 year
Reinfarction | 1 month
Major bleeding | during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Murat Sezer, M.D., Study Director — Istanbul University, Istanbul School of Medicine; Sabahattin Umman, Prof., Principal Investigator — Istanbul University, Istanbul School of Medicine; Taner Goren, Prof., Study Chair — Istanbul University, Istanbul School of Medicine; Huseyin Oflaz, Assoc.Prof., Study Chair — Istanbul University, Istanbul School of Medicine; Irem Okcular, M.D., Study Chair — Istanbul University, Istanbul School of Medicine; Yılmaz Nisanci, Prof., Study Chair — Istanbul University, Istanbul School of Medicine; Berrin Umman, Prof., Study Chair — Istanbul University, Istanbul School of Medicine; Ahmet K Bilge, M.D., Study Chair — Istanbul University, Istanbul School of Medicine; Mehmet Meric, Prof., Study Chair — Istanbul University, Istanbul School of Medicine
Locations (1):
- Istanbul University, Istanbul School of Medicine, Department of Cardiology, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Sezer M, Cimen A, Aslanger E, Elitok A, Umman B, Bugra Z, Yormaz E, Turkmen C, Adalet IS, Nisanci Y, Umman S. Effect of intracoronary streptokinase administered immediately after primary percutaneous coronary intervention on long-term left ventricular infarct size, volumes, and function. J Am Coll Cardiol. 2009 Sep 15;54(12):1065-71. doi: 10.1016/j.jacc.2009.04.083. PMID 19744615
- [Derived] Sezer M, Oflaz H, Goren T, Okcular I, Umman B, Nisanci Y, Bilge AK, Sanli Y, Meric M, Umman S. Intracoronary streptokinase after primary percutaneous coronary intervention. N Engl J Med. 2007 May 3;356(18):1823-34. doi: 10.1056/NEJMoa054374. PMID 17476008